CLINICAL TRIAL: NCT05721495
Title: Utility of Deferred Embryo Transfer in an In Vitro Program With Single Embryo Transfer Policy
Brief Title: Deferred Embryo Transfer in an In Vitro Program With Single Embryo Transfer Policy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Virgen de las Nieves (Other)
Collaborators: Junta de Andalucia (Other Government)
Responsible Party: Principal Investigator, Ana Clavero Gilabert, Medical Clinical laboratory especialist, University Hospital Virgen de las Nieves
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PI-0353-2016
Record Dates: First submitted 2022-12-16; First posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Single Embryo Transfer; Embryo Implantation, Delayed; Pregnancy Rate

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with two parallel arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study arm is masked until the oocyte recovery date, when we have to give a date in the control arm for the embryo transfer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Freeze all strategy embryo transfer (Experimental): Three days after fecundation, the best embryo is criopreserved. It is transferred in a posterior cicle
  Interventions: Other: freeze all strategy embryo transfer
- Fresh embryo transfer strategy (Active Comparator): Two or three days after fecundation, the best embryo is transferred.
  Interventions: Other: fresh embryo transfer strategy

INTERVENTIONS:
Other: freeze all strategy embryo transfer — criopreservation of all viable embryos in order to transfere the best one in a posterior cycle
  Arms: Freeze all strategy embryo transfer
Other: fresh embryo transfer strategy — transfer of the best embryo two or three days after the fecundation technique
  Arms: Fresh embryo transfer strategy

SUMMARY:
Single embryo transfer decreases the multiple pregnancy rate and its complications. However, studies are needed to help increase the effectiveness of this technique to increase its use, which undoubtedly improves the safety of our patients.

Objectives:

To assess the results of IVF / ICSI cycles with single embryo transfer, in terms of both pregnancy and live birth rates, comparing a group of patients in which an elective delayed cryotransfer of an embryo without fresh transfer is performed (experimental group ), with patients in whom a fresh embryo is transferred electively.

Methodology:

A prospective randomized clinical trial with two arms in parallel, not blinded, including 138 couples using an IVF / ICSI cycle at the Reproduction Unit of the Hospital Universitario Virgen de las Nieves de Granada. The inclusion criteria classify them as having a good reproductive prognosis, and the patients will follow an ovulation treatment protocol with GnRH agonists or antagonists. Couples will undergo an IVF / ICSI cycle, randomly assigned to:

* Group I (experimental): fresh transfer is not performed, the best quality embryo is cryopreserved. Elective transfer in a later cycle of the cryopreserved embryo.
* Group II (control): fresh transfer of the best quality embryo.

DETAILED DESCRIPTION:
The study has been designed as a prospective, randomized, two-arm, parallel, unblinded study, during which the investigators will include 138 couples (69 in each group) of IVF / ICSI users. Cycles canceled or punctured but without embryo transfer (either due to not obtaining oocytes, non-fertilization or arrest of embryonic development) will not be included in the study. The assignment of the couples to each of the groups will be carried out by means of a consecutive random sampling procedure. The randomization list will be created specifically for this project and will be kept safely by someone not included in the research team:

* Group I (experimental): fresh transfer is not performed, the best quality embryo is cryopreserved. Elective transfer in a later cycle of the cryopreserved embryo.
* Group II (control): fresh transfer of the best quality embryo.

Subjects of study:

Patients who come to the Human Reproduction Unit of the Virgen de las Nieves University Hospital to perform a first or second cycle of IVF / ICSI. Couples will be selected according to inclusion criteria that classify them as good reproductive prognosis (which is consistent with the usual eSET practice).

Couples will be able to participate in the study for only one cycle. Each couple will be interviewed to explain the characteristics of the study and will be given an Information Sheet. Written informed consent must be obtained from each couple. The person outside the research team who is guarding the randomization list will assign the corresponding treatment group.

Before starting the study, ethical approval was processed by the Ethics Committee through the Ethics Portal for Biomedical Research of Andalusia.

For the objective of assesing the null hypothesis that includes the equality of live birth rates in the group of women who undergo an elective deferred transfer of a single embryo and the group who undergo elective transfer of a fresh embryo, a power of 80% has been established to detect statistically significant differences by means of a bilateral Chi-square test for two independent samples, taking into account that the level of significance is 5%, and assuming that the proportion in the group of women who undergo a fresh transfer is 50.9%, the proportion in the group of women who receive the deferred elective transfer is 78%, and that the proportion of women with respect to the total is 50%, it will be necessary to include 48 women in each group, with the objetive to obtain 96 experimental units in the study. Taking into account that the expected dropout rate is three out of ten women, it will be necessary to include 69 women per group. The 138 women will be assigned to one of the groups using a random procedure, following a sequence of random numbers generated by specific software (Epidat, Epidemiological Data Analysis Program Tabulated. Version 3.1).

Methodology The patients must follow an ovulation stimulation treatment, in order to achieve multiple follicular development. A so-called "long analog" GnRH agonist protocol will be used. This consists of administering from day 22 of the cycle 0.1 mg / day of GnRH analog (Decapeptyl 0.1; Lasa, Barcelona, Spain) until the day on which the administration of gonadotropin is started, in which the dose is reduced at 50% until the day of hCG. After 10-14 days of administration of the agonist, the pituitary restraint is checked by means of ovarian vaginal ultrasound (absence of follicles and cysts) and serum estradiol determination (<50 pg / mL). If this medical hypophysectomy is confirmed, 300 IU of recombinant FSH (FSHr) is administered per day (Gonal F, Serono, Madrid, Spain) for two days, and 150 IU of FSHr from the 3rd to the 7th day. On this day, ultrasound monitoring of follicular development and serum estradiol determination are performed in order to once again adjust the dose of rFSH to each patient. Once the follicular response is adequate (more than 3 ovarian follicles greater than 18 mm in diameter), ovulation is triggered using 6,500 IU of hCG (Ovitrelle, Merck, Darmstadt, Germany).

IVF / ICSI and embryo culture will then be performed. To perform sperm microinsemination (ICSI) it is necessary to remove the cumulus and radiated crown from the oocyte. To decumulate, the crown-oocyte cluster complex is submerged in a solution with 80 IU / mL of hyaluronidase (HYASE, IVF Science Scandinavia, Gothenburg, Sweden) for 10-20 seconds, aspirating the complex several times using a pasteur pipette. The microinsemination technique is performed under an inverted microscope with Eppendorf and Narishigue micromanipulators and microinjectors. In Vitro Fertilization (IVF) is performed in a five-well plate, depositing 0.5 mL of IVF medium (Vitrolife, Sweden) and 0.5 mL of Ovoil (Vitrolife, Sweden) in each well. Five cumulus are left per well and 100,000 sperm / mL are added. In both cases, the oocytes are cultured in a Thermo-Fisher incubator, within a morphokinetic platform (PrimoVision) that takes photographs of them every 5-10 minutes. The following days are evaluated for classification, choosing the one with the best implantation potential according to the division times measured by morphokinetics and the morphological criteria of the Spanish Association for the Study of Reproduction Biology (ASEBIR) reviewed in 2015.

The embryo transfer will be carried out in group 2 on the third day choosing the best embryo according to the previous criteria. In group 1, the embryos will be cryopreserved by vitrification, selecting the best one for delayed transfer. The commercial vitrification media (Medicult Vitrification, Denmark) and the storage device will be Cryoleaf (McGill Cryoleaf, Medicult, Denmark). All cryopreserved embryos will be stored in liquid nitrogen at -196ºC in storage cylinders (Air Liquide, France). The day before cryotransfer the embryo is devitrified, using the thawing kit (Medicult Warming, Denmark). At the end, the embryo is washed in G2 medium (Vitrolife), leaving it in culture until the next day, after evaluating the embryo quality and cryosurvival (percentage of lysed cells). The woman's endometrium is prepared by treatment with estradiol valerate and progesterone. On the day of cryotransfer, embryo quality is assessed again, with emphasis on embryo division. Cryotransfer is performed using the same technique as transfer.

Study limitations The project has been carried out taking into account the resources available in the Human Reproduction Unit of the University Hospital Virgen de las Nieves, and therefore there do not seem to be any limitations in this regard.

The study could be completed by performing a preimplantation genetic diagnosis to determine if there are embryonic genetic alterations prior to intrauterine transfer, but this technique is not yet performed in our Unit. Likewise, blastocyst transfer can increase pregnancy rates, but by increasing the cancellation rate of embryo transfer, so it is not routinely performed in our Unit.

ELIGIBILITY:
Inclusion Criteria:

* BMI 19-29 kg/m2
* AMH > 0.5 ng/mL
* FIV/ICSI cycle: first or second

Exclusion Criteria:

* uterus surgery
* endometriosis
* miscarriage >1
* REM < 1 million spz

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Live birth rate | 15 months
  Live birth rate after freeze-all or fresh embryo strategy in an Assisted Reproduction program

SECONDARY OUTCOMES:
Metaphase II rate | 1 month
  Number of oocytes in Metaphase II stage of the total oocytes obtained
Fertility rate | 1 month
  Number of fertilized oocytes of the toal oocytes obtained
Good embryo quality rate | 1 month
  Number of embryos A or B of the total embryos obtained
Survival to devitrification rate | 4 months
  Number of embryos that survive to devitrification
Gestation rate | 4 months
  Clinical gestation rate (positive beta-hCG and positive heartbeat on 7 gestational week )
Implantation rate | 4 months
  Implantation rate
Miscarriage rate | 4 months
  Miscarriage rate
Newborn weight | 15 months
  Weight in grames of the newborn
Adverse events rates | 15 months
  Number of adverse events after or during treatment of the total treatments

CONTACTS AND LOCATIONS:
Overall Officials: Ana Clavero-Gilabert, PhD, Principal Investigator — HU Virgen de las Nieves
Locations (1):
- University Hospital Virgen de las Nieves, Granada, Spain

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT05721495/Prot_SAP_000.pdf